CLINICAL TRIAL: NCT02745496
Title: Multiparametric Magnetic Resonance Imaging Characterization and Guided Biopsy of the Prostate in Men Suspected of Having Prostate Cancer
Brief Title: Advanced Magnetic Resonance Imaging (MRI) in Men With Suspected Prostate Cancer
Acronym: MULTIPROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government); Prostate Cancer UK (Other); Tayside Clinical Trials Unit (Unknown); Health Informatics Centre (Unknown); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Principal Investigator, Ghulam Nabi, Professor in Surgical Uro-oncology, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MULTIPROS Study
Record Dates: First submitted 2016-03-04; First posted 2016-04-20 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
Keywords: Image-guided biopsy; Tumour detection; Diagnostic; Biomarkers
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRUS Biopsy (Other): Standard of Care Treatment
  Interventions: Procedure: TRUS Biopsy
- TRUS/FUSION Biopsy (Other): Interventional Treatment
  Interventions: Procedure: TRUS/FUSION Biopsy

INTERVENTIONS:
Procedure: TRUS Biopsy — Standard of Care Treatment
  Arms: TRUS Biopsy
Procedure: TRUS/FUSION Biopsy — Interventional Treatment
  Arms: TRUS/FUSION Biopsy

SUMMARY:
The clinical trial aims to address the critical challenge of differentiating aggressive from indolent prostate cancers by correlating prospectively collected MultiParametric (MP) Magnetic Resonance Imaging (MRI) data (index test) with the histopathology of radical prostatectomy specimens (reference standard).

The study design incorporates pre-biopsy MRI, routine standard of care Transrectal Ultrasound guided (TRUS) biopsies and MRI/Ultrasound (US) image fusion techniques to guide biopsies to the suspicious areas identified by MRI.

The hypothesis is that MP-MRI will allow pre-treatment determination of prostate cancer aggressiveness and MRI/US image fusion is expected to accurately co-locate cancer foci within the prostate gland for guiding biopsies.

Pre-treatment prediction of Gleason grade as a marker of cancer aggressiveness will better inform clinicians and patients to improve risk stratification and facilitate decision making on subsequent treatment.

Image fusion will allow accurate targeting of the most suspicious areas on MP-MRI for biopsy, which could obviate the need for multiple biopsies.

DETAILED DESCRIPTION:
There is preliminary evidence suggesting that MultiParametric Magnetic Resonance Imaging (MP-MRI) can be a marker for prostate cancer (PCa) aggressiveness and could be used to plan treatment. Gleason grade (GG) is a critical predictor of the aggressiveness of PCa, but in up to one in three men, the histology of radical prostatectomy specimens is different from the histology of Transrectal Ultrasound (TRUS)-guided biopsies. This discrepancy contributes to- and is a sign of- poor risk stratification of men with localised PCa.

The research aims to answer the following questions:

1. Can image-fusion techniques allow investigators to reliably target abnormal areas seen on MP-MRI?
2. How reliable is pre-biopsy MP-MRI in correctly predicting aggressive disease?

The investigators envisage that MP-MRI information will reduce unnecessary biopsies and over-detection of indolent PCa, while improving the detection of aggressive disease.

Primary Objectives

• To determine whether using MP-MRI can improve cancer detection and characterization of prostate cancer

Secondary Objectives

• To determine whether US/MRI FUSION guided biopsy can reduce the number of false negative biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Males between the age of 40-75 at referral
* With at least 10 years life expectancy
* With clinically localised PCa: Prostate Specific Antigen (PSA) ≤20 ng/ml
* And/or abnormal Digital Rectal Examination (DRE) but < T3 disease
* Ability to informed consent

Exclusion Criteria:

* Unable to give informed consent
* Prior prostatic biopsy within 12 months
* Contraindications to biopsy
* Poor general health and life expectancy < 10 years
* Previous diagnosis of acute prostatitis within 12 months
* History of prostate cancer
* Prior transurethral prostatectomy
* Contraindications to MRI (cardiac pacemakers, allergic reaction to gadolinium based contrast, renal function with baseline eGRF 30 ml/min, intracranial clips, claustrophobia)
* Previous hip replacement

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Number of prostate cancers detected by MP-MRI when compared to gold standard prostatectomy specimen | 5 years from first recruitment
  Number of prostate cancers detected by MP-MRI when compared to gold standard
Number of clinically significant cancers detected by MP-MRI when compared to gold standard prostatectomy specimen | 5 years from first recruitment
  The definition of clinically significant disease will be based on the pathologic assessment of radical prostatectomy (RP) specimen and will include the presence of any the following three prognostic factors:
  o Gleason grade >= 7 with pattern 4 or/and 5 Maximum cancer focus size more than 6mm measured in the axial plane Presence of extracapsular extension (ECE)

SECONDARY OUTCOMES:
Number of cancer detected in each randomised group, namely intervention group (TRUS/FUSION biopsy) versus standard of care (TRUS biopsy) | 5 years from first recruitment
  Number of cancer detected in each randomised group
Number of significant cancer detected in each randomised group, namely intervention group (TRUS/FUSION biopsy) versus standard of care (TRUS biopsy) | 5 years from first recruitment
  Number of significant cancer detected in each randomised group
Safety outcomes(death, post biopsy pain, bleeding, sepsis and hospitalization) of intervention (biopsy) in each of the two randomised groups. | 4 years from first recruitment
  Number of participants with deaths, side effects (post biopsy pain, bleeding, sepsis and hospitalization) in each of the two randomised groups.
Comparison of MRI negative standard of care TRUS guided biopsies with MRI positive TRUS histopathology to facilitate analysis of diagnostic accuracy of MRI in men suspected with target condition. | 5 years from first recruitment
  Comparison of MRI negative standard of care TRUS guided biopsies with MRI positive TRUS histopathology

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Nabi, Study Director — University of Dundee
Locations (1):
- Ninewells Hospital and Medical School, Dundee, Tayside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei C, Szewczyk-Bieda M, Bates AS, Donnan PT, Rauchhaus P, Gandy S, Ragupathy SKA, Singh P, Coll K, Serhan J, Wilson J, Nabi G. Multicenter Randomized Trial Assessing MRI and Image-guided Biopsy for Suspected Prostate Cancer: The MULTIPROS Study. Radiology. 2023 Jul;308(1):e221428. doi: 10.1148/radiol.221428. PMID 37489992
- [Derived] Szewczyk-Bieda M, Wei C, Coll K, Gandy S, Donnan P, Ragupathy SKA, Singh P, Wilson J, Nabi G. A multicentre parallel-group randomised trial assessing multiparametric MRI characterisation and image-guided biopsy of prostate in men suspected of having prostate cancer: MULTIPROS study protocol. Trials. 2019 Nov 21;20(1):638. doi: 10.1186/s13063-019-3746-0. PMID 31752954